CLINICAL TRIAL: NCT02467790
Title: Kinetic Study of Human Pharmacokinetics in Normal Renal Function, and Renal Insufficiency Subject of Polyethylene Glycol Loxenatide (PEX168)(Open, Non-randomized, Parallel-group)
Brief Title: Polyethylene Glycol Loxenatide Pharmacokinetics Study in Subjects With Normal and Insufficiency Renal Function
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEX168-Ih
Record Dates: First submitted 2015-06-08; First posted 2015-06-10 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — polyethylene glycol loxenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mild renal insufficiency (Experimental): PEX 168: 200µg,Subcutaneous,one time.
  Interventions: Drug: PEX168
- Moderate renal insufficiency (Experimental): PEX 168: 200µg,Subcutaneous,one time.
  Interventions: Drug: PEX168
- Normal renal function (Experimental): PEX 168: 200µg,Subcutaneous,one time.
  Interventions: Drug: PEX168

INTERVENTIONS:
Drug: PEX168 — PEX 168: 200µg,Subcutaneous,one time.
  Other Names: Polyethylene Glycol Loxenatide

SUMMARY:
To compare and analysis pharmacokinetics of PEX 168 in patients with renal insufficiency or normal renal function who were administrated subcutaneously single dose PEX168.To evaluate dose adjustment of PEX168 administered in patients with renal insufficiency and provide a scientific basis in patients with renal insufficiency of rational drug use.

DETAILED DESCRIPTION:
This is an open, non-randomized, parallel-group, single-dose study that evaluated the pharmacokinetics of PEX168 when single dose administered with PEX168 in patients with renal insufficiency and normal renal function subjects. The total duration of each subject's participation in the study was approximately 45 days, which included up to a 14-day Screening Period, a 31-day PK sample collecting Period.

Center: This study was conducted at two sites in the Third Xiangya hospital of Center South University and Shanghai Changhai Hospital.All subjects receives a single 200μg doses of PEX168 injected subcutaneously on Day 1.

ELIGIBILITY:
Inclusion Criteria:

1. Age 31-65 (both inclusive) years old, male or female;
2. Weight: Male ≥50kg, female ≥45kg, 18≤BMI≤28;
3. The Cockcroft-Gault (CG) formula to estimate creatinine clearance (CLCr), K / DOQI definition of chronic kidney disease (CKD) 2 patients: 60≤CLcr≤89 ml / min; chronic kidney disease (CKD) 3 patients: 30≤CLcr≤59 ml / min for renal insufficiency,Cockcroft-Gault (CG) formula to estimate creatinine clearance (CLCr) ≥90ml / min for normal subjects.
4. In the 48 hours before the start of the test to the end of the trial period, agreed to get rid of tobacco, alcohol, caffeine, fruit juice subject;
5. Understand the study procedures and methods, voluntarily participate in this experiment, and writing and signed informed consent.

Exclusion Criteria:

1. Known or suspected of GLP-1 class of drug allergy or allergy;
2. Before screening,received GLP-1 receptor agonists, GLP-1 analogs, DPP-IV inhibitors or any other similar structure of the drug treatment;
3. In addition to the induced renal dysfunction disease itself, suffering from any other organ of acute illness and those with any influence of drugs in vivo study of chronic diseases;
4. within 6 months prior to screening,having any surgery, including the impact of gastric emptying of gastrointestinal surgery;
5. Screened within the previous three months to participate in blood donation and blood donation ≥400mL, or who participate in blood donation or blood transfusion within one month;
6. Within 3 months before screening participated in any drug or medical device trials are (including placebo);
7. Drinking, smoking addiction, drug abuse and drug abusers;
8. In addition to judging laboratory abnormalities diagnosis of renal dysfunction caused by disease, there are other clinically significant laboratory abnormalities (Note: Patients with moderate to severe anemia (Hb <60g / L), severe hypertension ( SBP> 160mmHg and / or diastolic blood pressure> 100mmHg) patients, heart rate> 100bmp, ECG QTc> 450ms were required to exclude;
9. ALT> 1.5 times the upper limit of normal and / or aspartate transaminase> 1.5 times the upper limit of normal and / or total bilirubin> 1.5 times the upper limit of normal;
10. Fasting triglycerides> 5.64mmol / L (500mg / dl);
11. Beyond the normal range of serum amylase, and the clinical significance is determined by the investigator;
12. Pancreatitis, pancreatic cancer a history;
13. Blood thyroid stimulating hormone (TSH) beyond the normal range and clinically significant judgment by the investigator;
14. The pregnancy test was positive women of childbearing age, or pregnant women, breastfeeding women, and within six months there have been unwilling or unable to take family planning and effective contraception during the trial of male / female volunteers;
15. The hepatitis B surface antigen, hepatitis C antibody, HIV antibody, syphilis antibody test positive;
16. Researchers believe any situation that might lead to any subject can not be completed or to the subject of this study bring significant risk.

Ages: 31 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-03 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic index | Baseline to Day31
  Prior to administration (within 60 minutes, recorded as 0h) and after administration 24h (Day 2), 48h (Day 3), 72h (day 4), 96h (day 5), 120h (day 6 ), 144h (day 7), 216h (day 10), 312h (day 14 ), 480h (day 21), 648h (day 28), 720h (day 31) collect blood 3 ml and test serum concentrations of PEX168.

SECONDARY OUTCOMES:
Incidence of adverse events and serious adverse events | Baseline to Day31

CONTACTS AND LOCATIONS:
Overall Officials: Guoping Yang, MD, Principal Investigator — The Third Xiangya Hospital,Center South University
Locations (1):
- Third Xiangya Hospital, Central South Univety, Changsha, Hunan, China

REFERENCES:
- [Derived] Wang J, Huang J, Li W, Tang S, Sun J, Zhang X, Liu J, Yi B, Liu J, Zhang X, Yang Q, Yang X, Yang S, Yang G, Zhang H. Polyethylene glycol loxenatide (PEX168) in subjects with renal impairment: A pharmacokinetic study. Br J Clin Pharmacol. 2019 Dec;85(12):2714-2720. doi: 10.1111/bcp.14091. Epub 2019 Dec 8. PMID 31396983